CLINICAL TRIAL: NCT05615974
Title: A Phase I/II, Open-label, Dose Escalation, and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy of LM-101 Injection as a Single Agent or Combination Therapy in Patients With Advanced Malignant Tumors
Brief Title: A Phase I/II Study of LM-101 Injection in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM101-01-103
Record Dates: First submitted 2022-10-18; First posted 2022-11-14 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Malignant Tumors
MeSH Terms: conditions — Neoplasms | interventions — toripalimab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LM101 Dose Escalation (Experimental)
  Interventions: Drug: LM101
- LM101 combination therapy exploratory (Experimental)
  Interventions: Drug: LM101; Drug: Toripalimab; Drug: Rituximab
- LM101 combination expansion (Experimental)
  Interventions: Drug: LM101; Drug: Toripalimab; Drug: Rituximab

INTERVENTIONS:
Drug: LM101 — Administered intravenously
Drug: Toripalimab — Administered intravenously
  Arms: LM101 combination expansion; LM101 combination therapy exploratory
Drug: Rituximab — Administered intravenously
  Arms: LM101 combination expansion; LM101 combination therapy exploratory

SUMMARY:
This study is to assess the safety and tolerability, obtain Maximum Tolerated Dose (MTD) and/or the recommended phase 2 dose (RP2D) of LM-101 as a single agent or in combination in patients with advanced malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Aged ≥18 years old, male or female.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Life expectancy ≥ 3 months.
5. Subjects must have histological or cytological confirmation of recurrent or refractory advanced solid tumors, and have progressed on standard therapy.
6. At least one evaluable lesion.
7. Subjects in the combination therapy group must have Archived Samples or fresh tumor tissue specimens are required for testing.
8. Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose:
9. Women of childbearing potential (WOCBP) must agree to use highly effective methods of contraception prior to study entry, during the study and for 6 months after the last dose of study drug.
10. Subjects who can communicate well with investigators and understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Subject has received prior investigational therapy directed at the same target therapy.
2. Subjects has participated in any other interventional clinical trial within 21 days prior to the first dosing of LM-101.
3. Subjects with anti-tumor treatment within 21 days prior to the first dosing of LM-101, including radiotherapy, chemotherapy, endocrine therapy, and immunotherapy, etc.
4. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
5. Poorly controlled tumor-related pain.
6. Subjects with symptomatic/active central nervous system (CNS) metastases.
7. Subjects who have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
8. Subjects with known hypersensitivity to antibody therapy.
9. Subjects who take systemic corticosteroids (> 10 mg daily prednisone equivalents) or other systemic immunosuppressive medicationswithin 2 weeks prior to the first dosing of LM-101.
10. Subjects with the known history of autoimmune disease with the exception of subjects with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone.
11. Subject who has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
12. Use of any live attenuated vaccines within 28 days prior to the first dosing of LM-101.
13. Subjects who are using therapeutic doses of anticoagulants such as heparin or vitamin K antagonists.
14. Subjects who received major surgery or interventional treatment within 28 days prior to the first dosing of LM-101 (excluding tumor biopsy, puncture, etc.).
15. Subjects who have history of severe cardiovascular disease.
16. Subjects who have uncontrolled or severe illness.
17. Subjects who have a history of immunodeficiency disease.
18. HIV infection, active tuberculosis or active HBV and HCV infection.
19. Subjects who have Known history of active tuberculosis.
20. Subjects who have other active invasive cancers, other than the one treated in this trial, within 5 years prior to screening.
21. Child-bearing potential female who have positive results in pregnancy test or are lactating.
22. Subject who have a known psychiatric diseases or disorders that may affect compliance with the trial.
23. Subject who is judged as not eligible to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2028-01-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 48 weeks
  Phase 1
Incidence of dose-limitingtoxicity (DLT) | 48 weeks
  Phase 1
Incidence of serious adverse event (SAE) | 48 weeks
  Phase 1
Temperature in ℃ | 48 weeks
  Phase 1
Pulse in BPM(Beat per Minute) | 48 weeks
  Phase 1
Blood Pressure in mmHg | 48 weeks
  Phase 1
Weight in Kg | 48 weeks
  Phase 1
Height in centimeter | 48 weeks
  Phase 1
Laboratory tests-Blood Routine examination | 48 weeks
  Phase 1
Laboratory tests-Urine Routine test | 48 weeks
  Phase 1
Laboratory tests-Blood biochemistry | 48 weeks
  Phase 1
Laboratory tests- Coangulation function | 48 weeks
  Phase 1
Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage | 48 weeks
  Phase 1
12-lead electrocardiogram (ECG) in QTcF. | 48 weeks
  Phase 1
12-lead electrocardiogram (ECG) in QT. | 48 weeks
  Phase 1
12-lead electrocardiogram (ECG) in QRS. | 48 weeks
  Phase 1
12-lead electrocardiogram (ECG) in HR. | 48 weeks
  Phase 1
12-lead electrocardiogram (ECG) in RR. | 48 weeks
  Phase 1
12-lead electrocardiogram (ECG) in PR. | 48 weeks
  Phase 1
ECOG(Eastern Cooperative Oncology Group) score | 48 weeks
  Phase 1
Overall Response Rate (ORR) | 64 weeks
  Phase 2

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) | 112 weeks
  Phase 1 and 2
PK Parameter:Time of Maximum Observed Concentration (Tmax) | 112 weeks
  Phase 1 and 2
PK Parameter: Area Under the Concentration-time Curve(AUC) | 112 weeks
  Phase 1 and 2
PK Parameter: Steady State Maximum Concentration(Cmax,ss) | 112 weeks
  Phase 1 and 2
PK Parameter: Steady State Minimum Concentration(Cmin,ss) | 112 weeks
  Phase 1 and 2
PK Parameter: Systemic Clearance at Steady State (CLss) | 112 weeks
  Phase 1 and 2
PK Parameter: Accumulation Ratio (Rac) | 48 weeks
  Phase 1 and 2
PK Parameter: Elimination Half-life (t1/2) | 112 weeks
  Phase 1
PK Parameter: Volume of Distribution at Steady-State (Vss) | 112 weeks
  Phase 1 and 2
PK Parameter: Degree of Fluctuation (DF) | 112 weeks
  Phase 1 and 2
Immunogenicity of LM-101 | 112 weeks
  Phase 1 and 2; Anti-Drug antibody and Nab (if neccessary) will be tested.
Receptor Occupancy of LM-101 | 48 weeks
  Phase 1
Biomarker correlation (CD8/CD47/CD68/CD163/PD-L1) | 112 weeks
  Phase 1 and 2
Duration of Response (DOR) in Month | 64 weeks
  Phase 2
Disease control rate (DCR) in percentage | 64 weeks
  Phase 2
progression-free survival (PFS) in Month | 64 weeks
  Phase 2
Overall survival (OS) in Month | 64 weeks
  Phase 2
Changes of target lesions from baseline in Millimeter. | 64 weeks
  Phase 2
Safety: AE/SAE (Number of participants with treatment-related adverse events as assessed by CTCAE v5.0) | 64 weeks
  Phase 2
Temperature in ℃ | 64 weeks
  Phase 2
Pulse in BPM(Beat per Minute) | 64 weeks
  Phase 2
Blood Pressure in mmHg | 64 weeks
  Phase 2
Weight in Kg | 64 weeks
  Phase 2
Height in centimeter | 64 weeks
  Phase 2
Laboratory tests-Blood Routine examination | 64 weeks
  Phase 2
Laboratory tests-Urine Routine test | 64 weeks
  Phase 2
Laboratory tests-Blood biochemistry | 64 weeks
  Phase 2
Laboratory tests- Coangulation function | 64 weeks
  Phase 2
12-lead electrocardiogram (ECG) in RR, PR, QRS, QT, QTcF etc. | 64 weeks
  Phase 2
ECOG(Eastern Cooperative Oncology Group) score | 64 weeks
  Phase 2

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Linyi Cancer Hospital, Linyi, Shandong
  - Beijing Tongren Hospital, CMU, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No